CLINICAL TRIAL: NCT05293444
Title: Effect of Preoperative Carbohydrate Loading on Post-operative Insulin Resistance After Donor Hepatectomy: A Randomized Controlled Trial
Brief Title: Effect of Preoperative Carbohydrate Loading on Post-operative Insulin Resistance After Donor Hepatectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ILBS-Donor Hepatectomy-01
Record Dates: First submitted 2022-02-25; First posted 2022-03-24 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Overnight fasting (Other): overnight fasting(minimum 6 hrs) for control group.
  Interventions: Other: overnight fasting
- Maltodextrin (Experimental): Route: Oral Dose:
  * 400 ml at 10PM night before surgery(12.5g/100ml)
  * 200 ml in the morning at 6 AM (12.5g/100ml) on the day of surgery.
  Interventions: Dietary Supplement: Maltodextrine

INTERVENTIONS:
Dietary Supplement: Maltodextrine — 400 ml at 10PM night before surgery(12.5g/100ml) 200 ml in the morning at 6 AM (12.5g/100ml) on the day of surgery.
  Arms: Maltodextrin
Other: overnight fasting — no intervention
  Arms: Overnight fasting

SUMMARY:
It's a randomized control trial to compare the effect of preoperative carbohydrate loading versus fasting on post operative insulin resistance after donor hepatectomy in terms of donor outcomes. Investigator will analyze the data and elucidate the value of post operative insulin resistance in reducing the occurrence of complications, length of hospital stay and fastening the recovery in donors of Live donor liver transplantation.

DETAILED DESCRIPTION:
AIM: Investigator aim to study the effect of preoperative carbohydrate loading on insulin resistance and functional recovery after donor hepatectomy.

(B) Methodology: Present study will be a Randomized Control Trial with randomization into either study group or control group. Study group will undergo preoperative carbohydrate loading while control group will have conventional preoperative fasting (minimum 6 hours) in donors undergoing donor hepatectomy in live donor liver transplantation. Patients will be allocated to each arm on the basis of block randomization.

400 ml of clear carbohydrate drink (12.5 g/100 ml maltodextrin,50 kcal/100 ml) at 10 PM night before surgery & 200 ml, 2 hr before induction of anaesthesia will be given to the study group while overnight fasting(minimum 6 hrs) will be given for control group.

After donor hepatectomy, Insulin resistance will be calculated by HOMA-IR score at 6 AM on Day of Surgery, 6hrs after surgery, 12 hours and 36 hours (POD 2) after surgery. C-reactive protein and IL-6 at 6 AM on Day of Surgery, 48 hrs & on day 7 after surgery. Functional recovery of remnant liver will be assesed by normalization of total bilirubin and PT/INR till discharge and on day 14 after surgery. Peak lactate levels & time taken for normalization of lactate will be taken. Incidence of post operative nausea and vomiting and length of hospital stay will be compared between the two groups

Clinical and demographic parameters to be assessed- Donor-preoperative-Age, sex, BMI, LFTs, HbA1c, HOMA-IR, IL-6, CRP Operative parameters-duration of surgery, blood loss Postoperative serial measurements of the following parameters-

HOMA-IR, IL-6, CRP, Lactate level, LFTs, PT-INR, Post operative nausea & vomiting, Day of discharge These patients would be followed closely in the post-operative period and would be serially sampled at pre-defined time points for the aforementioned variables. At the end of the study the incidence of complications as well as improvement in postoperative recovery will be compared between the 2 groups. The clinical and laboratory parameters will be compared between those received preoperative carbohydrate loading and overnight fasting group.

Study Population: Consecutive patients undergoing live donor hepatectomy at ILBS during the study period.

Study Design:-Randomised Controlled Trial Study Period: December 2021 to May 2023. Inclusion Criteria All consecutive live liver donors who undergo donor hepatectomy at ILBS Exclusion criteria Patients refusing to consent for inclusion in the study. Donor hepatectomy for ALF(acute liver failure) recipient

Sample Size Assuming that HOMA-IR in conventional group is 1.7±0.1 and further investigator assume that there will be 25% reduction by preoperative carbohydrate loading with α-5%, Power- 90% and 1:1 ratio. Investigator need to enroll 70 cases i.e, 35 in each group. They will be randomly allocated in two groups by block randomization method, taking block size as 10 (5 in interventional & conventional group each).

Intervention: In Experimental group the preoperative carbohydrate loading will be done.

The control group will undergo overnight fasting (minimum 6 hrs) preoperatively.

Monitoring and Assessment:

Variables to be measured:

Donor- Preoperative parameters: age, sex, BMI, LFTs, HbA1c, HOMA-IR, IL-6, CRP Operative parameters: Duration of surgery, blood loss, Postoperative serial measurements of the following from day one to discharge HOMA-IR, Lactate, IL-6, CRP, LFTs, PT-INR, Post operative nausea & vomiting,

Day of discharge.

Timing of Sample Collection Group A Preoperative Baseline ( at 6 AM on day of surgery. Post-Operative:-6 hours after surgery & then daily till discharge. Group B Preoperative Baseline ( at 6 AM on day of surgery. Post-Operative:-6 hours after surgery & then daily till discharge. Adverse Effects: None

Statistical Analysis:

Data will be entered in excel worksheet and Statistical analyses will be performed with SPSS Statistics version 22 (IBM Corp., Armonk, NY). Statistical data will be represented as frequencies (%) where the continuous variables will be expressed as medians and interquartile range (IQRs). Continuous variables will be compared with the student t test and Mann-Whitney test as appropriate. Differences between proportions derived from categorical data will be compared with Chi-square or Fisher's exact test. Variables will be correlated with clinical outcomes. Repeated analysis of measures will be applied wherever applicable.

Stopping Rule- In case of significant adverse effects in the experimental arm. (c) EXPECTED OUTCOME:

1. To establish that preoperative carbohydrate loading will decrease the post operative insulin resistance and enhances functional recovery after donor hepatectomy.
2. To establish that preoperative carbohydrate loading reduces inflammatory stress response, incidence of post operative nausea & vomiting and improves the surgical clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive live liver donors who undergo donor hepatectomy at ILBS

Exclusion Criteria:

1. Patients refusing to consent for inclusion in the study.
2. Donor hepatectomy for ALF(acute liver failure) recipient

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
To compare the insulin resistance by HOMA-IR(Homeostatic model assessment for insulin resistance) on postoperative day 2 between preoperative carbohydrate loading and conventional fasting group after donor hepatectomy. | Post operative day 2

SECONDARY OUTCOMES:
To compare the functional recovery by total bilirubin on postoperative day 1 | Post operative day 1
To compare the functional recovery by PT/INR on postoperative day 1 | Post operative day 1
To compare the functional recovery by total bilirubin on postoperative day 3. | Post operative day 3
To compare the functional recovery by PT/INR on postoperative day 3. | Post operative day 3
To compare the functional recovery by total bilirubin on postoperative day 5. | Post operative day 5
To compare the functional recovery by PT/INR on postoperative day 5. | Post operative day 5
To compare the functional recovery by total bilirubin on postoperative day 7 | Post operative day 7
To compare the functional recovery by PT/INR on postoperative day 7 | Post operative day 7
To compare the functional recovery by total bilirubin on postoperative day 14. | Post operative day 14.
To compare the functional recovery by PT/INR on postoperative day 14. | Post operative day 14.
To compare the IL-6 levels after 48 hours of surgery. | 48 hours after surgery.
To compare the C-reactive protein levels after 48 hours of surgery. | 48 hours after surgery.
To compare the IL-6 levels on day 7 after surgery. | On day 7 after surgery.
To compare the C-reactive protein levels on day 7 after surgery. | On day 7 after surgery.
To compare the incidence of post operative nausea & vomiting till discharge | 1 week after surgery.
To compare the length of hospital stay. | 2 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Viniyendra Pamecha, MS, FRCS(UK), Study Director — Institute of Liver and Biliary Sciences, New Delhi
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, India

REFERENCES:
- [Derived] Kumar M, Patil NS, Mohapatra N, Yadav A, Sindwani G, Dhingra U, Thomas S, Pamecha V. Preoperative carbohydrate loading reduces perioperative insulin resistance and hastens functional recovery of remnant liver after living donor hepatectomy: An open-label randomized controlled trial. Hepatol Int. 2025 Oct;19(5):1151-1161. doi: 10.1007/s12072-025-10831-5. Epub 2025 May 19. PMID 40389625